CLINICAL TRIAL: NCT02526758
Title: Evaluation and Treatment of Small Airways in COPD
Brief Title: Small Airways Evaluation and Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SACOPD2015
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Disease，Chronic Obstructive;
Keywords: Pulmonary disease; chronic obstructive; small airway
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Beclomethasone; Formoterol Fumarate; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- beclomethasone / formoterol (Experimental): beclomethasone 100ug and formoterol 6ug , 2 inhalations, twice daily ,for three months
  Interventions: Drug: beclomethasone; Drug: formoterol
- budesonide / formoterol (Active Comparator): budesonide 160ug and formoterol 4.5ug, 2 inhalations ,twice daily ,for three month
  Interventions: Drug: formoterol; Drug: budesonide

INTERVENTIONS:
Drug: beclomethasone
  Other Names: Beclomethasone Dipropionate,BDP
  Arms: beclomethasone / formoterol
Drug: formoterol
Drug: budesonide
  Arms: budesonide / formoterol

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common disease , and characterized by progressive development of airflow limitation. Small airway disease (obstructive bronchitis) and lung parenchyma damage (emphysema) are the main mechanisms of chronic airflow limitation. Research shows that small airway resistance increased by 4-40 times in COPD patients, and become the main part of the airflow obstruction. Impulse oscillation system (IOS) is able to measure the total airway resistance, the central airway resistance and the peripheral airway resistance, which is now widely used to assess small airway function in COPD patients. While High resolution CT (HRCT) is easy to operate and its images are intuitive. Meanwhile it can measure the proportion of emphysema, the airway diameter and the thickness of airway wall. Both of these two tests have great significance in small airway evaluation. Chronic obstructive pulmonary disease with acute exacerbation (AECOPD) is an acute onset process, which is characterized by the aggravation of respiratory symptoms and deterioration of pulmonary function. However, the structural and functional changes of small airway in AECOPD are not clear. Inhalation drugs are the main treatment for stable COPD , and inhaled corticosteroid（ICS）+long-acting beta2-agonist（LABA） are used to treat patients with severe and severe airflow limitation. The particles in traditional inhalation drugs are larger and mainly deposited in large airways, and their effects on small airway function are relatively small.

The objectives of the investigators study are COPD patients. The study is divided into two parts, that is the part of AECOPD patients and the part of stable patients . Patients with AECOPD are arranged to take HRCT and IOS test to assess the small airway changes.Patients with stable COPD are randomized to take either beclomethasone / formoterol (particle diameter for 1.4-1.5um) or budesonide / formoterol (3.2um) for three months. The structure and function changes of small airway in different stage will be evaluated and the efficacy of these two drugs is to be compared. This study is expected to highlight the investigators understanding on the role of small airways in COPD, and provide a guideline to clinical standardized treatment as well as evaluation of patients' conditions.

DETAILED DESCRIPTION:
The COPD patients in the investigators hospital are selected to participate in the investigators study, and strict inclusion and exclusion criteria are to be complied with. All the subjects will be told the details of the study and sign the informed consent before inclusion.HRCT will be used to evaluate the structure of small airway by measuring the thickness of the third stage branches of apical segmental bronchus in the right upper lobe (WT). R5-R20 measured by IOS will be used to assess small airway resistance.

The study is divided into two parts, that is the part of AECOPD patients and the part of stable patients . Both of them have three steps .

Part 1. AECOPD patients:

* Subjects screening : To inquire the history of the disease and to take the IOS and Bronchial dilation test.
* Baseline data collection：patients will be arranged to complete a series of questionnaires, as well as HRCT, IOS, pulmonary function test and 6 minute walk test.
* Test stage：During their hospital stay, the patients are to be treated with oxygen inhalation and different kinds of drugs, and the patients will followed up for three weeks after discharge. Completing the examinations and questionnaires at each time visit ,and another CT scan at the last visit.

Part 2. Stable COPD patients:

* Subjects screening : To inquire the history of the disease and to take the IOS and Bronchial dilation test.
* Baseline data collection：In the two-week washout period，patients are only allowed take salmeterol/fluticasone 50:250ug 2 times daily, and stop the use of other inhalation drugs and oral glucocorticoid. At the end of this period, complete a series of questionnaires, as well as HRCT, IOS, pulmonary function test and 6 minute walk test.
* Test stage： patients are randomized to take either beclomethasone / formoterol (100:6ug 2inhalations twice daily ) or budesonide / formoterol (160:4.5ug 2inhalations twice daily) for three months.Completing the examinations and questionnaires at the end of each month, another CT scan at the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease;
* More than 40 years;

Exclusion Criteria:

* asthma , or combined with bronchiectasia，pneumonia in the right upper lobe;
* Malignant tumor in the lung or other parts of the body;
* Uncontrolled hypertension (systolic blood pressure >200 mmHg, diastolic blood pressure >100 mmHg);
* Severe cardiac insufficiency, arrhythmia;

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
R5-R20 measured by IOS | three month
  Change of small airway resistance (R5-R20)measured by IOS at three months

SECONDARY OUTCOMES:
forced expiratory volume at one second（FEV1） | three month
  change of forced expiratory volume at one second（FEV1） measured by pulmonary function test（PFT）at three months
Score of symptoms using the St. George respiratory questionnaire | three month
  The St. George respiratory questionnaire
Score of symptoms using modified Medical Research Council Dyspnoea Scale(mMRC) | three month
  modified Medical Research Council Dyspnoea Scale(mMRC)
Score of symptoms | three month
  CAT
Change of wall thickness（WT） | three month
  change of thickness of the third stage branches of apical segmental bronchus in the right upper lobe (WT) in three months

CONTACTS AND LOCATIONS:
Overall Officials: Huizhen Fan, Doctor, Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China